CLINICAL TRIAL: NCT02747641
Title: Prospective, Open-Label, Single-Center, Non-Comparative Study to Assess the Use of Pixel CO2 Laser System (FemiLift) in the Treatment of Vulvovaginal Atrophy (VVA) in Postmenopausal Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLA 15-110
Record Dates: First submitted 2016-04-12; First posted 2016-04-22 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2016-10

CONDITIONS: Atrophy; Vaginal Atrophy; Genital Diseases, Female
MeSH Terms: conditions — Atrophy; Genital Diseases, Female

ARMS (1):
- treatment (Other): only one arm
  Interventions: Procedure: Pixel CO2 Laser System

INTERVENTIONS:
Procedure: Pixel CO2 Laser System
  Other Names: FemiLift

SUMMARY:
The purpose of this study is to assess the use of the Alma CO2 Pixel FemiLift™ in the treatment of VulvoVaginal Atrophy (VVA) in postmenopausal female subjects. The primary endpoint is to assess the change in the vaginal dryness by means of a Visual Analogic Scale (10 cm VAS) and/or Bachmann Index in VVA. The clinical improvement will be assessed by patient filled Vulvovaginal Atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking
* Woman, age 35 to 70 yrs, menopausal
* Provided written Informed Consent
* Exhibiting VVA and/or SUI symptoms (mild or moderate SUI, according to severity index developed by Sandvik.)
* Prolapse staged < II, according to the pelvic organ prolapse quantification (ICS-POP-Q) system
* Normal PAP smear (up to 1 year prior to baseline)
* Vaginal canal, introitus and vestibule free of injuries and bleeding
* Have not had procedures in the anatomical area through 6 months prior to treatment
* Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

* Severe prolapse (POP>= grade 3)
* Use of photosensitive drugs
* Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. herpes candida).
* Any serious disease, or chronic condition, that could interfere with the study compliance
* Acute or actively present within the last 2 months HPV/HSV
* Undiagnosed vaginal bleeding
* Urge or overflow incontinence
* Patients who are on antidepressants, or α-adrenergic and anticholinergic medications
* Patients with immune system diseases.
* Patients with allergic reaction to laser.
* Obese women (BMI >30)
* Patient unable to follow post-treatment instructions
* History of keloid formation
* Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti inflammatories within 2 weeks pre treatment
* A history of thrombophlebitis
* A history of acute infections
* A history of heart failure
* Previously undergone reconstructive pelvic surgery
* Have used vaginal creams, moisturizers, lubricants or homeopathic preparations for at least 3 months
* Any medical condition that in the investigators opinion would interfere with the patients participation in the study

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Vulvovaginal Atrophy (VVA) | 6 months
  Utilizing Bachman Vaginal Health Index

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic, Weston, Florida, United States